CLINICAL TRIAL: NCT03952572
Title: Open-label Multi-center Randomized Non-inferiority Study to Compare Efficacy and Safety of Pegylated Liposomal Doxorubicin Versus Doxorubicin for Newly Diagnosed Peripheral T-cell Lymphoma
Brief Title: Efficacy and Safety of CDOP vs CHOP for Newly Diagnosed Peripheral T-cell Lymphoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Jun Zhu, Principal Investigator, Peking University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-DMS-LY-02
Record Dates: First submitted 2019-05-10; First posted 2019-05-16 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Peripheral T-cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — Cyclophosphamide; liposomal doxorubicin; 1-dodecylpyridoxal; Vincristine; Prednisone; Doxorubicin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CDOP regimen (Experimental): cyclophosphamide, pegylated liposomal doxorubicin, vincristine and prednisone (CDOP) administered in 3 week cycles for 6 cycles.
  Interventions: Drug: Cyclophosphamide; Drug: pegylated liposomal doxorubicin; Drug: Vincristine; Drug: Prednisone
- CHOP regimen (Active Comparator): cyclophosphamide, doxorubicin, vincristine and prednisone (CHOP) administered in 3 week cycles for 6 cycles.
  Interventions: Drug: Cyclophosphamide; Drug: Vincristine; Drug: Prednisone; Drug: Doxorubicin

INTERVENTIONS:
Drug: Cyclophosphamide — 750mg/m² ivgtt on day 1
  Other Names: CTX
Drug: pegylated liposomal doxorubicin — 40mg/m² ivgtt on day 1
  Other Names: PLD
  Arms: CDOP regimen
Drug: Vincristine — 1.4mg/m²(Maximum 2 mg) ivgtt on day 1
  Other Names: VCR
Drug: Prednisone — Prednisone100mg/m² po on day1-5
  Other Names: PED
Drug: Doxorubicin — 50mg/m² ivgtt on day 1
  Other Names: DOX
  Arms: CHOP regimen

SUMMARY:
Primary objective of the study is to compare the efficacy and safety of CDOP versus CHOP for newly diagnosed peripheral T-cell lymphoma (PTCL).

DETAILED DESCRIPTION:
This is a open-label, multi-center, randomized, non-inferiority study to compare efficacy and safety of CDOP with standard CHOP regimen in patients with previously untreated PTCL. Study subjects are patients with histologically proven newly diagnosed PTCL. Patients are randomized 1:1 to receive either cyclophosphamide, pegylated liposomal doxorubicin, vincristine and prednisone (CDOP) administered in 3 week cycles for 6 cycles or cyclophosphamide, doxorubicin, vincristine and prednisone (CHOP) administered in 3 week cycles for 6 cycles.This study is divided into three phases: screening phase, treatment phase and follow-up phase. Patients will receive study drug(s) for up to 6 cycles, or until unacceptable toxicity will develop or progression or voluntary withdrawal.Adverse event of every treatment cycle will be recorded.Therapy efficacy will be evaluated after finishing 2 cycles, 4cycles and finishing 6 cycles therapy. Patients will be followed until disease progression, died or 2 years from the last patient randomized.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically proven untreated peripheral T-cell lymphoma (include PTCL not otherwise specified（PTCL-NOS）, angioimmunoblastic T cell lymphoma（AITL）, anaplastic large cell lymphoma（ALCL）and other peripheral T-cell lymphoma(except NK/T cell lymphoma);
2. Males and females of 18 years of age to 75 years of age.
3. Eastern Cooperative Oncology Group (ECOG) performance status 0- 2.
4. At least 1 single size measurable lesions, CT or PET-CT scan shows more than 15mm.
5. Estimated survival time ≥ 6 months
6. Liver function: transaminases≤3×ULN，or transaminases≤3×ULN for liver metastasis，total bilirubin ≤1.5ULN，or total bilirubin ≤2.5ULN for Gilbert's syndrome
7. Renal function: serum creatinine ≤1.5×ULN or creatinine clearance ≥ 60 ml / min ( standard Cockcroft-Gault formula);
8. peripheral hemogram: WBC≥3.0×10^9/L, ANC≥1.5×10^9/L, Hb≥90g/L, PLT≥75×10^12/L.
9. Cardiac ultrasound LVEF≥55%;
10. New York Heart Association (NYHA) heart function classification is I grade;
11. sign informed consent.

Exclusion Criteria:

1. Patients with primary or secondary central nervous system lymphoma；
2. Serious heart disease, including but not limited to:

1)Significant ventricular arrhythmia or high degree atrioventricular block (Mobitz II or third degree atrioventricular block); 2) unstable angina; 3) clinically significant heart valve disease; 4) Electrocardiogram shows transmural myocardial infarction; 5) Uncontrollable hypertension; 3. interstitial pneumonia, allergic asthma or severe allergic medical history; 4.Patients with other malignancies in the past or now (except basal cell carcinoma, squamous-cell carcinoma or carcinoma in situs of cervix that has been adequately treated), 5.HIV antibody positivity; 6.Acute or chronic active hepatitis B (HBsAg positivity, HBV DNA negative acceptable), acute or chronic active hepatitis C (HCV antibody negatively acceptable; HCV antibody positivity, HCV RNA negative acceptable) 7.Pregnancy or lactation period 8.Patients with Organ transplantation 9.Patients with serious uncontroled acute infection 10.High doses of hormones are contraindicated, such as uncontrolled hyperglycemia, stomach ulcers or Mental illness, etc.

11.Patients with severe neurological or psychiatric history, including dementia or epilepsy 12.The researchers considered that patients are not suitable for the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Estimated)
Dates: Start 2019-05-10 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Response rate | 2 years
  complete response (CR) and partial response (PR) rates, using the standard response criteria

SECONDARY OUTCOMES:
Progression Free Survival | 2 years
  from date of inclusion to date of progression, relapse, or death from any cause
Overall Survival | 2 years
  from the date of inclusion to date of death, irrespective of cause
Cardiac toxicity | 2 years
  cardiotoxity Congestive heart failure with clinical symptoms, or no symptoms but an abnormal LVEF
Adverse Events | 2 years
  any unfavorable and unintended sign , symptom, or disease temporally associated with the use of a medical treatment or procedure that may or may not be considered related to the medical treatment or procedure

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhu, PHD, Study Chair — Peking University Cancer Hospital & Institute
Locations (1):
- Peking University Cancer Hospital & Institute, Beijing, Beijing Municipality, China